CLINICAL TRIAL: NCT02250729
Title: Anaphylaxis to Neuromuscular Blocking Agents and Pholcodine Exposure. Case-control Study
Brief Title: Allergy to Neuromuscular Blocking Agents and Pholcodine Exposure
Acronym: ALPHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Zambon SpA (Industry); Laboratoires URGO (Industry); THE BOOTS COMPANY PLC (Unknown); Pierre Fabre Medicament (Industry); LABORATOIRE HEPATOUM (Unknown); Biocodex (Industry); Sanofi (Industry); RECORDATI GROUP (Industry); GlaxoSmithKline (Industry); ALLIANCE PHARMACEUTICALS LIMITED (Unknown); BELL SONS & COMPANY (Unknown); PINEWOOD LABORATORIES LIMITED (Unknown); THORNTON & ROSS & Ross Ltd (Unknown); ERNEST JACKSON & Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A01735-38
Record Dates: First submitted 2014-05-12; First posted 2014-09-26 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Neuromuscular Blocking Agents Anaphylaxis
Keywords: anaphylaxis; pholcodine; neuromuscular blocking agents
MeSH Terms: conditions — Anaphylaxis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cases with NMBA anaphylaxis (Experimental): Patients who experienced NMBA anaphylaxis during anesthesia
  Interventions: Other: intradermal pholcodine allergy test in cases; Other: Blood sampling
- controls (Other): Patients who underwent anesthesia with NMBA injection but did not experience anaphylaxis
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: intradermal pholcodine allergy test in cases
  Arms: cases with NMBA anaphylaxis
Other: Blood sampling

SUMMARY:
The main objective of this study is to compare pholcodine exposure in patients having presented with a perianaesthetic anaphylactic reaction to a NMBA (cases) to pholcodine exposure in matched anaesthetised patients with injection of NMBA, who did not present with an anaphylactic reaction (controls).

The secondary objectives of the study are:

* To compare anti-pholcodine IgE, anti-ammonium IV IgE and total IgE levels between the case and control groups.
* To study the concordance between exposure to pholcodine in cases and controls, by means of a patient self-questionnaire on the one hand and, on the other hand, by a computerized drug history, supplemented where relevant by the drug master file.
* To study the impact of taking 1, 2 or 3 sources in account for pholcodine exposition.
* To study the association between exposure to pholcodine and the presence/levels of pholcodine-specific IgE, reflecting sensitisation to pholcodine.
* To study NMBA and pholcodine cross-sensitisation by testing skin reactions to pholcodine in case patients allergic to (at least) one NMBA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 2 years old.
* Referred to anaesthesia-allergy consultation within (approximately) 6 to 12 weeks of occurrence of peranaesthetic anaphylactic reaction during anaesthesia with administration of NMBAs (only for case patient).
* Having given his/her consent (or the 2 parents consent for minors).
* Affiliated with a social security scheme or dependent.
* Able to answer a medicinal product intake questionnaire
* In a clinical condition compatible with skin tests (no skin disease or psychiatric illness, etc.) (only for case patient)
* Having stopped any anti-histamine treatment at least 8 days previously (only for case patient).
* With positive skin test for the suspected NMBA (ony for case patient).
* Patient anaesthetised in a control recruitment centre (only for control patients)
* Having undergone anaesthesia with NMBA injection, without onset of peranaesthetic anaphylactic reaction whatever his medical history (only for control patients)

Exclusion Criteria:

* Patients who have refused, or are unable to give their consent
* Patients who have had negative control skin tests
* Anaphylaxis suspected to be related to other drugs given on induction of anaesthesia, eg. antibiotics
* Having presented with anaphylactic reaction during a previous anaesthesia without NMBA injection
* Pregnant females at inclusion or during 12 months before anaesthesia

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Exposure to pholcodine | within the 12 months before the anesthetic procedure
  Exposure is measured by autoquestionnaire, patient's pharmaceutical file and drug history by the pharmacist's

SECONDARY OUTCOMES:
Anti-pholcodine IgE, anti-ammonium IV IgE and total IgE levels between the case and control groups. | Between 1 day to 12 weeks after the general anesthetic procedure
  Cases: 6 to 12 weeks after the general anesthetic procedure (corresponding to the day of inclusion) Controls: during their hospitalisation after the general anesthetic procedure (Maximum 90 days after the general anesthetic procedure, corresponding to the day of inclusion)
Concordance between exposure to pholcodine in cases and controls, by means of a patient self-questionnaire on the one hand and, on the other hand, by a computerized drug history, supplemented where relevant by the drug master file. | within the 12 months preceeding the general anesthesia
Impact of non subjective sources in pholcodine exposure assessment | within the 12 months preceeding general anesthetic procedure
  We will study if pholcodine exposure criteria measured by autoquestionnaire is modified by taking into account non subjectives sources which are the patient's pharmaceutical file and his drug history by his pharmacist's
Association between exposure to pholcodine and the presence/levels of pholcodine-specific IgE, reflecting sensitisation to pholcodine. | within the 12 months preceding the general anesthetic procedure
  IgE measurements: total IgE, IgE specific for pholcodine, quaternary ammoniums (KU/L)
NMBA and pholcodine cross-sensitisation by testing skin reactions to pholcodine in case patients allergic to one NMBA. | 6 to 12 weeks after the general anesthetic procedure
  Only for Cases :
  Intradermal tests with diluted pholcodine. Intradermal tests with diluted NMBAs (as usual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GILLET, PU-PH MD, Principal Investigator — Central Hospital, Nancy, France; Paul-Michel MERTES, PU-PH MD, Study Director — CHU de Strasbourg
Locations (24):
- France (24):
  - CHU d' ANGERS, Angers
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - AP-HM, Marseille
  - CHU de MONTPELLIER, Montpellier
  - CHRU de Nancy, Nancy
  - CHU de NANTES, Nantes
  - CHU de Nice, Nice
  - Fondation Hôpital St Joseph, Paris
  - AP-HP- Hôpital Bichat, Paris
  - AP-HP Paris TENON, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU de Rouen, Rouen
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de TOURS, Tours

REFERENCES:
- [Derived] Mertes PM, Petitpain N, Tacquard C, Delpuech M, Baumann C, Malinovsky JM, Longrois D, Gouel-Cheron A, Le Quang D, Demoly P, Gueant JL, Gillet P; ALPHO Study Group. Pholcodine exposure increases the risk of perioperative anaphylaxis to neuromuscular blocking agents: the ALPHO case-control study. Br J Anaesth. 2023 Jul;131(1):150-158. doi: 10.1016/j.bja.2023.02.026. Epub 2023 Mar 24. PMID 36967281